CLINICAL TRIAL: NCT05251285
Title: Post Market Clinical Follow-up Study on da Vinci® Robotic-assisted Prophylactic Nipple Sparing Mastectomy With Breast Reconstruction
Acronym: PREVENT
Status: Terminated | Type: Observational
Why Stopped: Low enrolment
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: PN #1082409C
Record Dates: First submitted 2022-02-02; First posted 2022-02-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Prophylactic Nipple Sparing Mastectomy (NSM)
Keywords: robot; robotic; Nipple Sparing Mastectomy; NSM; da Vinci; surgery; mastectomy; prophylactic NSM; robot-assisted
MeSH Terms: interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prophylactic Nipple-Sparing Mastectomy
  Interventions: Procedure: Nipple-Sparing Mastectomy

INTERVENTIONS:
Procedure: Nipple-Sparing Mastectomy — Nipple-Sparing Mastectomy using da Vinci X/Xi Surgical System

SUMMARY:
The objective of this study is to collect post-market clinical safety and performance data on the robotic assisted prophylactic Nipple Sparing Mastectomy (R-NSM) surgery performed with the da Vinci Xi/X Surgical System as part of a PMCF Plan.

DETAILED DESCRIPTION:
This is an observational post-market study. Women will be screened for participation where the decision to undergo prophylactic R-NSM surgery has already been made as part of their medical care. In order for women to be enrolled, surgeons must perform the surgery according to the Instructions For Use (IFU) of da Vinci Xi/X Surgical System. Women will sign an informed consent form for their participation in the study. Women will be prospectively followed at 6 weeks, 3 months and 1 year post-surgery, which is within the standard of care. Data will be collected prospectively from the medical records and women will be asked to complete preoperative and postoperative questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a woman, candidate for a prophylactic R-NSM surgical procedure (unilateral or bilateral) according to the Instructions For Use (IFU) of da Vinci Xi/X Surgical System
* Subject has cup size A, B or C,
* Subject is 18 years of age or older,
* Subject is a candidate for reconstruction,
* Subject is willing to participate as demonstrated by signing the informed consent,
* Subject benefits from a health care system/insurance.

Exclusion Criteria:

* Subject is pregnant or is lactating,
* Subject has active cancer or pre-cancer (Ductal Carcinoma In Situ [DCIS]) on breast to be robotically operated,
* Subject has cancer involving the Nipple Areolar Complex (NAC), inflammatory breast cancer or T4d lesion, clinical evidence of skin involvement or T4b lesion, and clinical or radiological evidence of chest wall invasion.
* Subject has ASA score ˃ III or has known thromboembolism risks or, is at risk in relation to anesthesia,
* Subject presents severe lack of cooperation due to psychological or severe systemic illness,
* Subject has medical conditions contraindicating general anesthesia or surgical approach,
* Subject is part of vulnerable population (e.g., prisoners, mentally disabled).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women eligible for prophylactic robotic-assisted Nipple-Sparing Mastectomy (unilateral or bilateral) according to the Instructions For Use (IFU) of da Vinci Xi/X Surgical System
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Number of intraoperative R-NSM procedure and device-related complications | Assessed during surgery to 42 days after surgery
Number of overall post-operative complications at 6 weeks | 6 weeks after the surgery
Number of overall post-operative complications at 3 months | 3 months after the surgery
Number of overall post-operative complications at 1 year | 1 year after the surgery
Nipple-Areola Complex (NAC) necrosis occurrence (using SKIN composite score definition of D2 or higher) observed at 6 weeks after surgery | 6 weeks after surgery
Nipple-Areola Complex (NAC) Preservation Rate at 6 weeks after surgery | 6 weeks after surgery
Number of conversions to open surgery | Assessed during surgery
OR & procedure (open surgery dissection, docking and console) times, including drainage and reconstruction times | Assessed during surgery to 6 weeks after surgery
Number of transfusion and transfused units | Assessed during surgery to 6 weeks after surgery
Hospital Length of Stay (LOS) | Assessed during the 6 weeks after surgery
Results of the SKIN score (Mayo clinic) at 6 weeks or upon surgeon's practice | at 6 weeks or upon surgeon's practice
Number of readmissions associated with NSM surgery at 6 weeks | 6 weeks after surgery
Number of readmissions associated with NSM surgery at 3 months | 3 months after surgery
Number of reoperations associated with NSM surgery at 6 weeks | 6 weeks after surgery
Number of reoperations associated with NSM surgery at 3 months | 3 months after surgery
Result of BREAST-QTM (Quality of life) at 3 months | 3 months after surgery
Result of BREAST-QTM (Quality of life) at 1 year | 1 year after surgery
Result of NAC questionnaire (Quality of life) at 3 months | 3 months after surgery
Result of NAC questionnaire (Quality of life) at 1 year | 1 year after surgery
Breast Cancer Occurrence Assessment at 1 year according to usual medical practice | 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Toesca, MD, Principal Investigator — Istituto Europeo di Oncologia; Benjamin Sarfati, MD, Principal Investigator — Gustave Roussy Cancer Campus
Locations (2):
- Gustave Roussy Cancer Campus, Villejuif, France
- Istituto Europeo di Oncologia, Milan, Italy

IPD SHARING:
Plan to Share IPD: No